CLINICAL TRIAL: NCT01499498
Title: A Phase I Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of Boceprevir and Sildenafil When Dosed Separately and Together in Healthy Male Volunteers
Brief Title: The Boceprevir and Sildenafil Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOC_PK
Record Dates: First submitted 2011-11-04; First posted 2011-12-26 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C
Keywords: Healthy volunteers
MeSH Terms: conditions — Hepatitis C | interventions — Sildenafil Citrate; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sildenafil and Boceprevir (Experimental): Healthy volunteers
  Interventions: Drug: Sildenafil and Boceprevir

INTERVENTIONS:
Drug: Sildenafil and Boceprevir — 25mg once/800mg three times a day
  Other Names: Viagra and Victrelis

SUMMARY:
This is a healthy volunteer study looking at the interactions between two drugs: boceprevir and sildenafil.

New drugs are being developed to treat people with the chronic viral infection hepatitis C. Very little is know how these new treatments interact with other medications such as the drugs used to treat erectile dysfunction.

The purpose of this study is to look at levels of both a new hepatitis C drug called boceprevir (BOC) and an existing erectile dysfunction drug called sildenafil to see if they affect the blood levels of each other when given separately and together.

DETAILED DESCRIPTION:
Total duration for each participant will be up to 40 days plus a screening visit 1 - 3 weeks prior to the start of the study.

They will visit the clinic on 10 occasions: screening visit, baseline visit (day 0), day 1, a visit between day 4 and 7, day 10, day 14, day 15, day 16, day 17 and a follow up visit between days 26 and 40.

The total amount of blood collected from participants during the entire study will be no greater than 350 ml in total (around 23 tablespoons).

At the screening visit a clinical assessment will be performed. At the baseline visit participants will attend the clinic fasted and will be required to remain on the unit for approximately 14 hours.

On the morning of the visit clinical assessments will be performed. Sildenafil 25mg (1 tablet) will be administered with a standardised meal. Blood samples will be taken at the following times in order to measure the levels of sildenafil in the blood: predose,0.5, 1, 2, 3, 4, 6, 8, 10,12 and 24 hours post dose.

On day Day 10 boceprevir will be initiated 800mg (4 capsules 3 times a day) for the next 4 days on day 14 the participants will attend the clinic for a witnessed dose of boceprevir and safety assessment.

On day 15 the participants will attend for their 2nd long visit (10 hours) when they will be administered boceprevir (BOC) 800mg (4 capsules) with a standardised meal then have blood samples taken at the following times in order to measure the levels of BOC in the blood: predose,0.5, 1, 2, 3, 4, 6 and 8 hours post dose.

After the 8 hour blood collection participants will be administered boceprevir (BOC) 800mg (4 capsules) with food and they will self administer BOC 800mg (4 capsules) with food at home 8 hours later.

On day 16 participants will attend for the 3rd long visit (14 hours) where they will be administered boceprevir (BOC) 800mg (4 capsules) and sildenafil 25mg with a standardised meal. Blood samples will be taken at the following times in order to measure the levels of both BOC and sildenafil in the blood: predose,0.5, 1, 2, 3, 4, 6 and 8 hours post dose.

After the 8 hour blood collection participants will be administered boceprevir (BOC) 800mg (4 capsules) with food and will then self administer BOC 800mg (4 capsules) with food at home 8 hours later. This will be their last dose of study medication. They will return the next day for a final blood test post 24 hours. A final visit between days 26 and 40 will be performed including clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.
* Subjects in good health upon medical history, physical exam, and laboratory testing and BMI <32.
* Subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom with spermicide) during heterosexual intercourse, from screening through completion of the study including 10 days following last dose of study drug.
* Have no serologic evidence of HIV or HCV infection through antibody testing at screening.
* Have screening laboratory results (haematology, chemistry) that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical relevance

Exclusion Criteria:

* Any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic (thyroid disorders, adrenal disease), immunodeficiency disorders, active infection, or malignancy.
* Previous participation in an investigational trial involving administration of any investigational compound within 1 month prior to the study screening.
* Clinically relevant alcohol or drug use (positive drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
* Any medication taken listed in protocol including over-the-counter medications and herbal products within 21 days of commencing study drug dosing with the exception of vitamins and/or paracetamol. When a concomitant medication is necessary, this will be reviewed by the Investigator and if not contraindicated, may be continued at the same dose and frequency during the study period.
* History of drug sensitivity or drug allergy which in the opinion of the investigator may put the subject at increased risk of drug reactions during the study.
* Subjects with female partners who are pregnant will not be allowed to enter the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MBChB MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil and Boceprevir: Healthy volunteers
  Sildenafil and Boceprevir : 25mg once daily/800mg three times a day
Period: Overall Study
Arm/Group | Sildenafil and Boceprevir
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil and Boceprevir: All subjects take single dose sildenafil 25mg day 0, day 10-15 they take boceprevir 800mg three times a day followed by Intentive PK on day 15 and on day 16 single dose of sildenafil and boceprevir together followed by intensive PK
Arm/Group | Sildenafil and Boceprevir
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 36 [22 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Median (Full Range); unit: kg/m2] | 26.2 [19.9 to 30.6]

OUTCOME MEASURES:

1. Primary Outcome: Sildenafil Alone Maximum Plasma Concentration
Description: Single dose sildenafil 25mg will be administered with food. Intensive pharmacokinetic sampling will be taken over a 24 hour period (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose)
Time Frame: Day 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Sildenafil Only: Healthy volunteers
  Sildenafil 25mg once
Arm/Group | Sildenafil Only
Number analyzed (Participants) | 13
ng/mL | 79.9 [59.9 to 106.5]

2. Primary Outcome: Boceprevir Alone Maximum Plasma Concentration
Description: Day 10 commence BOC 800mg three times a day with food. On day 15 at steady state, subjects will attend for witnessed dosing and an intensive pharmacokinetic visit over 8 hours (samples drawn 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post dose)
Time Frame: day 10-15
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Bocepreprivir Alone: Healthy volunteers
  Boceprevir: 800mg three times a day
Arm/Group | Bocepreprivir Alone
Number analyzed (Participants) | 13
ng/mL | 1432.5 [1276.1 to 1607.7]

3. Primary Outcome: Sildenafil Maximum Plasma Concentration
Description: administer BOC 800mg and single dose sildenafil 25mg with food. Intensive pharmacokinetic sampling will be taken over a 24 hour period (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post dose)
Time Frame: Day 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sildenafil and Boceprevir
Number analyzed (Participants) | 13
ng/mL | 150.9 [126.2 to 180.5]

4. Primary Outcome: Boceprevir Maximum Plasma Concentration
Description: as for outcome 3
Time Frame: Day 16
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Sildenafil and Boceprevir
Number analyzed (Participants) | 13
ng/mL | 1440.5 [1211.7 to 1712.4]

5. Secondary Outcome: Number of Patients With Adverse Events
Description: The number of repeated adverse events will be used to assess the safety of the drugs in combination
Time Frame: Day 1 - 16
Measure: Number; unit: participants
Arm/Group | Sildenafil and Boceprevir
Number analyzed (Participants) | 13
participants | 0

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | Sildenafil and Boceprevir
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No